CLINICAL TRIAL: NCT01340560
Title: The Effect of Local Injury to the Endometrium for Implantation and Pregnancy Rates in ICSI -ET Cycles With Recurrent Implantation Failure: a Randomised Controlled Study
Brief Title: Endometrial Injury Increases Implantation and Pregnancy Rates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Selcuk University Meram Medical Faculty
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: ref.no:2008-274
Record Dates: First submitted 2011-04-13; First posted 2011-04-22 (Estimated); Last update posted 2011-04-22 (Estimated); Status verified 2011-04

CONDITIONS: Focus of Study Instead
Keywords: Endometrium, local injury, implantation, pregnancy, in vitro fertilization

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Endometrial biopsy — Endometrial biopsy was performed with biopsy catheter

SUMMARY:
Objective To evaluate the effect of local injury to the endometrium for implantation, pregnancy and live birth rates in ICSI -ET cycles with recurrent implantation failure.

Design Randomized controlled clinical study. Setting A clinical will assist reproductive center of Selcuk University Meram Medical Faculty Hospital in the Konya, Turkey.

Population A group of 100 women, who failed to conceive during one or more cycles of IVF and embryo transfer (ET), will treat with a long protocol for controlled ovarian hyperstimulation.

Methods The IVF treatment and ET will precede by repeated endometrial biopsies, in a randomly selected 50 of a total of 100 women.

DETAILED DESCRIPTION:
The clinical study will take place in clinical assisted reproductive center of Selcuk University Meram Medical Faculty Hospital in the Konya, Turkey. A group of 100 women who apply to our clinic due to infertility and who undergo one or more failed fresh IVF cycles previously will be included in our study for ICSI-ET (intracytoplasmic sperm injection-embryo transfer).

We will exclude women with factors as hydrosalpinx, trombophilia, submucous myoma and found to have a negative impact on implantation. Women will be given information about the study, and written informed consents will be obtained. Our study also received approval of ethic committee of our faculty.

Women of the study group (n=50) will randomly selected. The random allocation will base on computer generated random numbers. All 100 women will treate with long protocol for COH (control group=group 1, n=50 and study group=group 2, n=50.

On the other hand, the women in the study group (group 2, n=50) will undergo endometrial biopsies with one-week intervals at the luteal phase of nontransfer cycle. Endometrial biopsy will performe with biopsy catheter (Pipelle; de Cornier, Prodimed, Neuilly-en-Thelle, France). The catheter will be passed through the cervical os and will rotate in uterine cavity and apply 3-4 times after withdrawing the piston.

Treatment schedules Administration of Leuprolide acetate (Lucrin; Abbott, France) at a subcutaneous dose of 1 mg/day will be started at the 21st day of menstrual cycle on the patient selected for therapy. All of the women will be protected by one of non-hormonal contraception method during this cycle.

After administration of GnRH analog at 2nd-3rd day of next menstruation or at least for 14 days in women without menstruation, patients with criteria including serum estrogen (E2) level is below 50 pg/ml, endometrial thickness is <5mm, lack of observation of active follicle on transvaginal ultrasonography will be accepted as down regulation, and gonadotropin therapy [recFSH; Puregon (Organon), Gonal F (Serono), u-FSH/HMG; Merional (IBSA), Menogon (Ferring)] will be started at a properly adjusted dose for each patient. Estimated ovarian response will be considered for each case while determining initial dose. While starting SC/I.M. gonadotropin of average dose 225 IU/day, GnRH analog (Leuprolide acetate; Lucrin, Abbott) will be maintained until hCG day by reducing to 0.5 mg/day doze uninterruptedly. When leading follicle will become 18-20 mm or two of follicles will become 17 mm, ovulation will be triggered by administering 10.000 IU urinary hCG (Pregnyl amp; Organon, Turkey).

Follicle aspiration and oocyte collection procedure will be performed at the range of 35th-37th hours following hCG administration.

Semen specimens will be collected on the day when follicle aspiration will be performed several hours before the procedure by masturbation method generally after sexual fasting of 2-4 days. Sperms of total 6 men, equally 3 men from each group, will be obtained by TESA/TESE method.

Microinjection procedure into suitable and adequate number of oocytes will be performed following oocyte collection procedure. Development of fertilized oocytes will be followed up under suitable laboratory conditions in culture dish (5% CO2, 95% humidity, 37º C temperature). Fertilization rates will be evaluated at the subsequent 18th hour and embryo development will be evaluated at 24th-48th-72nd hours. On 2nd-3rd or 4th day following oocyte collection, maximum 3 embryos having highest quality scores (grade 3 or 4 embryos will be considered to be good quality embryos) will be selected, and will be transferred into intrauterine cavity with accompaniment of ultrasonography. Wallace 23 mm soft catheter (Smiths, England) will be used as transfer catheter. Follicle aspiration and embryo transfer procedures will be performed by same physician in our study.

Luteal phase support will be started at the evening of follicle aspiration on all women. Use of intravaginal micronized progesterone 3x200 mg (Progeston soft capsule; Kocak ilac, Turkey), intramuscular progesterone 25 mg/day (Progeston in oil), prednisol tablet for 5 days in 16 mg/ day p.o. dose (Mustafa Nevzat, Turkey) and Estraderm TTS 100 (Novartis Pharma, Basel, Switzerland) 100 microgram/ on alternate days will be recommended until pregnancy result became apparent.

ELIGIBILITY:
Inclusion Criteria:

* women who applied to our clinic due to infertility and who undergone one or more failed fresh IVF cycles previously has been included in our study for ICSI-ET (intracytoplasmic sperm injection-embryo transfer).

Exclusion Criteria:

* women with factors as hydrosalpenx, trombophilia, submucous myoma and found to have a negative impact on implantation

Ages: 25 Years to 36 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-01 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Implantation ratio | Six months
  Implantation ratios were 30.88% in Group 1 and 34.67% in Group 2 (p =0.13). So there wasn't any significant difference for implantation ratios between two groups, but implantation ratio of 34.67% in Group 2 was evaluated as clinically significant
Clinical pregnancy ratio | six months
  Cardiac activity on USG for clinical pregnancy were determined in seventeen women of the control group (34%) and 30 women of the study group (60%). The clinical pregnancy rate was significiantly higher in the study group with compared to control group (p=0.009)
Live birth ratio | six months
  Twenty two of the 30 pregnancies in the study group ended in the delivery of 27 healthy babies. This stituation represents a rate of live births in the study group that was significiantly higher than control group (44% and 24%) (p= 0.03)

SECONDARY OUTCOMES:
Implantation ratio | six months
  Implantation ratios were 30.88% in Group 1 and 34.67% in Group 2 (p =0.13). So there wasn't any significant difference for implantation ratios between two groups, but implantation ratio of 34.67% in Group 2 was evaluated as clinically significant
Clinical pregnancy ratio | six months
  Cardiac activity on USG for clinical pregnancy were determined in seventeen women of the control group (34%) and 30 women of the study group (60%). The clinical pregnancy rate was significiantly higher in the study group with compared to control group (p=0.009)
Live birth ratio | six months
  Twenty two of the 30 pregnancies in the study group ended in the delivery of 27 healthy babies. This stituation represents a rate of live births in the study group that was significiantly higher than control group (44% and 24%) (p= 0.03)

CONTACTS AND LOCATIONS:
Locations (1):
- IVF Unit, Department of Obstetrics and Gynecology, Selcuk University Meram Medical Faculty, Konya, Turkey (Türkiye)

REFERENCES:
- [Derived] Lensen SF, Armstrong S, Gibreel A, Nastri CO, Raine-Fenning N, Martins WP. Endometrial injury in women undergoing in vitro fertilisation (IVF). Cochrane Database Syst Rev. 2021 Jun 10;6(6):CD009517. doi: 10.1002/14651858.CD009517.pub4. PMID 34110001
- See also: Selcuk University — http://www.selcuk.edu.tr